CLINICAL TRIAL: NCT00070018
Title: Evaluation of CHOP Plus Involved Field Radiotherapy Followed by Yttrium-90 Ibritumomab Tiuxetan for Stages I, IE, and Non-Bulky Stages II and IIE, CD20 Positive, High-Risk Localized, Aggressive Histologies of Non-Hodgkin Lymphoma, Phase II
Brief Title: S0313 Cyclophosphamide, Doxorubicin, Vincristine, Prednisone, and Radiation Therapy Followed By Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Stage I or Stage II Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000329864; U10CA032102 (NIH); S0313 (Other: SWOG)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult Burkitt lymphoma; anaplastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Radiotherapy; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHOP + RT + Zevalin (Experimental): Patients first receive 3 cycles (21 days each) of CHOP, consisting of: cyclophosphamide 750 mg/m^2 on day 1, doxorubicin 50 mg/m^2 on day 1, vincristine 1.4 mg/m^2 on day 1, and prednisone 100 mg on days 1-5. Patients receive 4000-5000 cGy of radiation therapy in 25 fractions, starting 3 weeks after completion of CHOP. 3-6 weeks after completing RT, patients receive Zevalin, which consists of: rituximab 250 mg/m^2 on days 1 and 7, 8 or 9; In-111 ibritumomab tiuxetan 5 mCi within 4 hours after rituximab on day 1; and Y-90 ibritumomab tiuxetan 0.4 mCi/kg within 4 hours after rituximab on day 7, 8 or 9.
  Interventions: Biological: rituximab; Drug: Cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy; Biological: Yttrium-90 ibritumomab tiuxetan; Biological: Indium-111 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab — 250 mg/m^2, as part of Zevalin regimen
Drug: Cyclophosphamide — 750 mg/m^2
Drug: doxorubicin hydrochloride — 50 mg/m^2
Drug: prednisone — 100 mg
Drug: vincristine sulfate — 1.4 mg/m^2
Radiation: radiation therapy — 4000-5000 cGy total
Biological: Yttrium-90 ibritumomab tiuxetan — 0.4 mCi/kg
Biological: Indium-111 ibritumomab tiuxetan — 5 mCi

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Monoclonal antibodies, such as rituximab and yttrium Y 90 ibritumomab tiuxetan, can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Combining chemotherapy with radiation therapy and monoclonal antibody therapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy and monoclonal antibody therapy works in treating patients with stage I or stage II non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 2-year progression-free survival of patients with aggressive high-risk stage I or IE or non-bulky stage II or IIE CD20-positive non-Hodgkin's lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone and radiotherapy followed by rituximab and yttrium Y 90 ibritumomab tiuxetan.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Chemotherapy: Patients receive CHOP chemotherapy comprising cyclophosphamide IV over 1-2 hours, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Radiotherapy: Beginning 3 weeks after the completion of CHOP chemotherapy, patients undergo radiotherapy once daily 5 days a week for 4-5 weeks.
* Monoclonal antibody therapy: Beginning 3-6 weeks after the completion of radiotherapy, patients receive rituximab IV followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients then undergo whole body imaging. If ibritumomab tiuxetan biodistribution is acceptable, patients receive rituximab IV and yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 7, 8, OR 9.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Diffuse large B-cell
  * Mantle cell
  * High-grade B-cell, Burkitt's, or Burkitt-like
  * Anaplastic large cell (B-cell phenotype only)
* Stage I, IE, or non-bulky* stage II or IIE disease by Ann Arbor classification

  * Patients who have bulky stage II or IIE disease are ineligible even if, after resection, the measurements are less than 10.0 cm NOTE: *Non-bulky disease defined as any tumor measuring less than 10.0 cm or occupying less than 1/3 of the chest diameter
* CD20-expressing disease by flow cytometry or immunoperoxidase staining
* Aggressive lymphomas must have at least 1 of the following adverse prognostic factors:

  * Non-bulky stage II or IIE disease
  * At least 60 years of age
  * Zubrod performance status of 2
  * Lactic dehydrogenase greater than upper limit of normal
* All disease must be encompassable in a single radiation port (including any site of resected disease) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No medical contraindication to study chemotherapy, rituximab, or ibritumomab tiuxetan
* No known AIDS syndrome or HIV-associated complex

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior monoclonal antibody therapy

Chemotherapy

* No prior chemotherapy for lymphoma

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy for lymphoma
* No concurrent intensity-modulated radiotherapy
* Planned involved-field radiotherapy must not encompass more than 25% of active bone marrow space

Surgery

* See Disease Characteristics

Other

* Concurrent participation in SWOG-8947 or SWOG-8819 allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-02; Primary Completion 2010-11 (Actual); Study Completion 2015-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Miller, MD, Study Chair — University of Arizona; Oliver W. Press, MD, PhD, Study Chair — Fred Hutchinson Cancer Center; Baldassarre D. Stea, MD, PhD, Study Chair — University of Arizona; Louis S. Constine, MD, Study Chair — James P. Wilmot Cancer Center
Locations (48):
- United States (48):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Miller TP, Unger JM, Spier C, et al.: Effect of adding ibritumomab tiuxetan (Zevalin) radioimmunotherapy consolidation to three cycles of CHOP plus involved-field radiotherapy for limited-stage aggressive diffuse B-cell lymphoma (SWOG 0313). [Abstract] Blood 112 (11): A-3598, 2008.
- [Derived] Persky DO, Miller TP, Unger JM, Spier CM, Puvvada S, Stea BD, Press OW, Constine LS, Barton KP, Friedberg JW, LeBlanc M, Fisher RI. Ibritumomab consolidation after 3 cycles of CHOP plus radiotherapy in high-risk limited-stage aggressive B-cell lymphoma: SWOG S0313. Blood. 2015 Jan 8;125(2):236-41. doi: 10.1182/blood-2014-06-584623. Epub 2014 Nov 13. PMID 25395425

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHOP + RT + Zevalin
Started | 46
Eligible | 46
Eligible and Began Protocol Therapy | 46
Completed | 42
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | CHOP + RT + Zevalin
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 61.2 [23.5 to 84.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 42
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Measured from date of registration to date of first observation of progression or symptomatic deterioration. Progression is defined as one or more of the following must occur. Unequivocal progression of disease in the opinion of the treating physician (an explanation must be provided). Appearance of a new lesion/site. Death due to disease without documented progression or symptomatic deterioration. Symptomatic deterioration is defined as global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: at 6 weeks after treatment, then every 6 months for 2 years, then annually thereafter
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHOP + RT + Zevalin
Number analyzed (Participants) | 46
percentage of participants | 89 [76 to 95]

ADVERSE EVENTS:
Time Frame: After each cycle of CHOP, after RT, and 3 months after Zevalin therapy for a maximum of 10 months
Arm/Group | CHOP + RT + Zevalin
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 44/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP + RT + Zevalin (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 28
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 10
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 6
Esophagitis (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 21
Pain - Oral cavity (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 11
Edema: limb (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 33
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 4
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3
Rash: dermatitis associated with radiation - Radiation (Injury, poisoning and procedural complications) | 16
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 8
Bilirubin (hyperbilirubinemia) (Investigations) | 3
Creatinine (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 29
Lymphopenia (Investigations) | 19
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 27
Platelets (Investigations) | 25
Weight loss (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 12
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 5
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Neuropathy: sensory (Nervous system disorders) | 14
Pain - Head/headache (Nervous system disorders) | 6
Taste alteration (dysgeusia) (Nervous system disorders) | 3
Mood alteration - depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 4
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 4
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 24
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No